CLINICAL TRIAL: NCT04683471
Title: Pilot Feasibility Clinical Validation Study
Brief Title: Pilot Trial of a System for Motor Function Recovery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Niche Biomedical, Inc. dba ANEUVO (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EXA-2001
Record Dates: First submitted 2020-12-15; First posted 2020-12-24 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Spinal Cord Diseases
MeSH Terms: conditions — Spinal Cord Diseases | interventions — Tissue Therapy, Historical

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Neuromodulation (Experimental): Neuromodulation
  Interventions: Device: Stimulator
- Sham (Sham Comparator): Sham
  Interventions: Device: Sham

INTERVENTIONS:
Device: Stimulator — Neuromodulation
  Arms: Neuromodulation
Device: Sham — Sham
  Arms: Sham

SUMMARY:
This is a multi-center, prospective, blinded, pilot feasibility study to evaluate improvement in sensory and motor function with sham.

ELIGIBILITY:
Inclusion Criteria:

* Traumatic chronic spinal cord injury

Exclusion Criteria:

* Active implanted medical device
* Internal metallic objects of unknown or foreign origin
* Implanted anti-spasticity pumps, Botox injections in prior 3 months or other current anti-spasticity regimen
* BMI > 40.0
* Acute medical conditions under active treatment that would contraindicate standard rehabilitation including open wounds
* Pregnancy or planned pregnancy
* Unhealed bone fractures, peripheral neuropathies or painful musculoskeletal dysfunction
* Cardiopulmonary disease or ventilator dependency
* Uncontrolled epilepsy or seizures
* Clinically significant depression, psychiatric disorders or ongoing substance abuse

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2021-12-22 (Actual); Study Completion 2022-03-22 (Actual)

PRIMARY OUTCOMES:
Graded Redefined Assessment of Strength, Sensibility and Prehension (GRASSP) | Biweekly through study completion up to 18 weeks
  Change in Graded Redefined Assessment of Strength, Sensibility and Prehension (GRASSP) for the upper limbs
  Scoring:
  * Strength scored 0 - 50 for each arm
  * Sensibility scored 0 - 24 for each arm
  * Prehension scored 0 - 42 for each arm
  * Higher scores are a better outcome

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Shirley Ryan AbilityLab, Chicago, Illinois
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Houston Methodist Research Institute, Houston, Texas